CLINICAL TRIAL: NCT03143088
Title: The Effect of Medical Clowns on Blood Pressure Measurement in Children Presenting to the Emergency Department
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, omer raviv, Principal Investigator, Meir Medical Center
Other Study IDs: MMC 034116 CTIL
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Children Referred to the Pediatric Emergency Department
Keywords: Blood pressure; Medical clown; Pediatric

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medical clown: Medical clown will be present in the pediatric emergency department while assessing blood pressure during triage of patients.
  Interventions: Behavioral: Medical clown
- Blood pressure assessment: Blood pressure will be measured by the medical center protocols.

INTERVENTIONS:
Behavioral: Medical clown — Blood pressure will be taken to children admitted to the pediatric emergency department with and without the presence of a medical clown.
  Groups: Medical clown

SUMMARY:
Obtaining vital signs and blood pressure (BP) in particularly, as part of a pediatric Emergency Department (ED) patient triage is sometimes difficult and leads to many false negative results.

The stress, noisy environment and lack of cooperation are only a few of the things that interfere with proper vital signs measurements.

In the past decade, there has been a rapid growth in the presence of therapeutic clowns in hospitals, particularly in pediatric settings.

The investigators speculate that the incorporation of a medical clown during the procedure of blood pressure measurement in the triage will shorten the procedure and decrease the number of attempts, making it much more efficient.

DETAILED DESCRIPTION:
Blood pressure is measured in the triage amongst most children presented to the Pediatric ED.

There are many barriers to obtaining an accurate BP measurement in children, including inappropriate technique, lack of equipment, but also - pain, and the child's uncooperativeness or anxiety. The latter may even be accentuated in an ED setting.

These factors may lead to falsely elevated BP readings, which may provoke significant anxiety in children and families and possibly lead to a cascade of unnecessary investigation and consultations.

Additionally, an abnormal measured BP value routinely mandate an additional measurement attempt which itself may cause anxiety and restlessness among children, especially toddlers and infants, and prolongs the entire triage process.

The Second Task Force Report on Blood Pressure Control in Children emphasizes taking blood pressure measurements in a quiet environment, using a proper size cuff and using appropriate technique. Ideally, BP should be measured several times in a a relaxed child and in a quiet setting, however this scenario is nearly impossible in the ED, as demonstrated in a previous retrospective study that indicated that although BP was elevated in 52% of children who underwent triage blood pressure measurement in the ED, the measurement was repeated in only 38%.

In the past decade, there has been a rapid growth in the presence of therapeutic clowns in hospitals, particularly in pediatric settings. A recent study conducted in a pediatric ED in Israel has demonstrated the benefit of medical clowns in diminishing pain and anxiety during painful procedures being performed on children in the ED.

Previous studies conducted in our institute have demonstrated a beneficial effect on vital signs (blood pressure and heart rate) as a sign of decreased anxiety following the incorporation of a medical clown in a multisystem team caring for pediatric patient.

Blood pressure measurement among pediatric patients, although not a painful procedure, may cause a stressful reaction, prolonging the entire process and requiring additional attempts - making it a time consuming task in a busy ED.

A medical clown may have a beneficial effect on the pediatric patient by decreasing the stress reaction and may therefore shorten the entire process making it much more efficient.

The investigators are unaware of any studies conducted related to the effect of the use of medical clowns during ED blood pressure measurements in the triage.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 day to 18 years presenting to the ED.

Exclusion Criteria:

1. Serious medical condition requiring emergent medical care or resuscitation
2. Parental refusal to participate in the study

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children population
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-08-06 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Accurate blood pressure assessment | 10 min
  Blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Omer Raviv, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Pediatrics Emergency Department, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No